CLINICAL TRIAL: NCT00364013
Title: A Randomized, Multicenter, Phase 3 Study to Compare the Efficacy of Panitumumab in Combination With Oxaliplatin/ 5-fluorouracil/ Leucovorin to the Efficacy of Oxaliplatin/ 5-fluorouracil/ Leucovorin Alone in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: PRIME: Panitumumab Randomized Trial In Combination With Chemotherapy for Metastatic Colorectal Cancer to Determine Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050203
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Oncology; Cancer; metastatic colorectal cancer; EGFr; Panitumumab; Clinical Trail; Amgen
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Panitumumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX + Panitumumab (Experimental): Participants received panitumumab, 6 mg/kg on Day 1 and FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Panitumumab; Drug: FOLFOX regimen
- FOLFOX (Active Comparator): Participants received FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or until unacceptable toxicity.
  Interventions: Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg over on Day 1 of each 14-day cycle, just prior to the administration of chemotherapy.
  Other Names: Vectibix®
  Arms: FOLFOX + Panitumumab
Drug: FOLFOX regimen — The FOLFOX regimen consisted of oxaliplatin 85 mg/m^2 intravenous (IV) infusion on Day 1, leucovorin, 200 mg/m^2 (racemate) on Days 1 and 2 and 5-fluorouracil 400 mg/m^2 IV bolus followed by 600 mg/m^2 IV infusion over 22 hours on Days 1 and 2. Each cycle was 14 days.

SUMMARY:
The purpose of this study is to determine the treatment effect of panitumumab in combination with FOLFOX compared to FOLFOX alone as first line therapy for metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Man or woman at least 18 years old
* Diagnosis of metastatic colorectal cancer
* At least 1 uni-dimensionally measurable lesion of at least 20 mm per modified RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Paraffin-embedded tumor tissue from the primary tumor or metastasis available for central analyse Exclusion Criteria:
* History or known presence of central nervous system (CNS) metastases
* History of another primary cancer, except: Curatively treated in situ cervical cancer, or Curatively resected non-melanoma skin cancer, or Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 5 years before randomization
* Prior chemotherapy or systemic therapy for the treatment of metastatic colorectal carcinoma except: adjuvant fluoropyrimidine-based chemotherapy or prior fluoropyrimidine therapy administered solely for the purpose of radiosensitization
* Prior oxaliplatin therapy
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (eg, cetuximab) or treatment with small molecule EGFr inhibitors (eg, erlotinib)
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 1 year prior to randomization History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > Common terminology criteria (CTC) grade 2 [CTCAE version 3.0])
* Peripheral sensory neuropathy with functional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1183 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2013-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Tian Y, Xu F, Sidhu R. Final results from PRIME: randomized phase III study of panitumumab with FOLFOX4 for first-line treatment of metastatic colorectal cancer. Ann Oncol. 2014 Jul;25(7):1346-1355. doi: 10.1093/annonc/mdu141. Epub 2014 Apr 8. PMID 24718886
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Background] Douillard JY, Siena S, Peeters M, Koukakis R, Terwey JH, Tabernero J. Impact of early tumour shrinkage and resection on outcomes in patients with wild-type RAS metastatic colorectal cancer. Eur J Cancer. 2015 Jul;51(10):1231-42. doi: 10.1016/j.ejca.2015.03.026. Epub 2015 May 5. PMID 25956209
- [Derived] Liu J, Wang X, Sahin IH, Imanirad I, Felder SI, Kim RD, Xie H. Tumor Response-speed Heterogeneity as a Novel Prognostic Factor in Patients With Metastatic Colorectal Cancer. Am J Clin Oncol. 2023 Feb 1;46(2):50-57. doi: 10.1097/COC.0000000000000972. Epub 2022 Dec 26. PMID 36606664
- [Derived] Taieb J, Geissler M, Rivera F, Karthaus M, Wilson R, Loupakis F, Price T, Tracy M, Burdon P, Peeters M. Relationship Between Tumor Response and Tumor-Related Symptoms in RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses From 3 Panitumumab Trials. Clin Colorectal Cancer. 2019 Dec;18(4):245-256.e5. doi: 10.1016/j.clcc.2019.07.009. Epub 2019 Jul 29. PMID 31515083
- [Derived] Abdel-Rahman O. Effect of Body Mass Index on 5-FU-Based Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer; A Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Dec;18(4):e385-e393. doi: 10.1016/j.clcc.2019.07.005. Epub 2019 Jul 15. PMID 31378656
- [Derived] Abdel-Rahman O. Impact of Sex on Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer: Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Jun;18(2):110-115.e2. doi: 10.1016/j.clcc.2018.12.006. Epub 2018 Dec 28. PMID 30679026
- [Derived] Modest DP, Rivera F, Bachet JB, de Braud F, Pietrantonio F, Koukakis R, Demonty G, Douillard JY. Panitumumab-based maintenance after oxaliplatin discontinuation in metastatic colorectal cancer: A retrospective analysis of two randomised trials. Int J Cancer. 2019 Jul 15;145(2):576-585. doi: 10.1002/ijc.32110. Epub 2019 Jan 24. PMID 30614531
- [Derived] Udar N, Lofton-Day C, Dong J, Vavrek D, Jung AS, Meier K, Iyer A, Slaughter R, Gutekunst K, Bach BA, Peeters M, Douillard JY. Clinical validation of the next-generation sequencing-based Extended RAS Panel assay using metastatic colorectal cancer patient samples from the phase 3 PRIME study. J Cancer Res Clin Oncol. 2018 Oct;144(10):2001-2010. doi: 10.1007/s00432-018-2688-3. Epub 2018 Jul 17. PMID 30019318
- [Derived] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Effect of Primary Tumor Location on Second- or Later-line Treatment Outcomes in Patients With RAS Wild-type Metastatic Colorectal Cancer and All Treatment Lines in Patients With RAS Mutations in Four Randomized Panitumumab Studies. Clin Colorectal Cancer. 2018 Sep;17(3):170-178.e3. doi: 10.1016/j.clcc.2018.03.005. Epub 2018 Mar 8. PMID 29627309
- [Derived] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Primary tumor sidedness has an impact on prognosis and treatment outcome in metastatic colorectal cancer: results from two randomized first-line panitumumab studies. Ann Oncol. 2017 Aug 1;28(8):1862-1868. doi: 10.1093/annonc/mdx119. PMID 28449055
- [Derived] Siena S, Tabernero J, Bodoky G, Cunningham D, Rivera F, Ruff P, Canon JL, Koukakis R, Demonty G, Hechmati G, Douillard JY. Quality of life during first-line FOLFOX4+/-panitumumab in RAS wild-type metastatic colorectal carcinoma: results from a randomised controlled trial. ESMO Open. 2016 Mar 31;1(2):e000041. doi: 10.1136/esmoopen-2016-000041. eCollection 2016. PMID 27843597
- [Derived] Peeters M, Kafatos G, Taylor A, Gastanaga VM, Oliner KS, Hechmati G, Terwey JH, van Krieken JH. Prevalence of RAS mutations and individual variation patterns among patients with metastatic colorectal cancer: A pooled analysis of randomised controlled trials. Eur J Cancer. 2015 Sep;51(13):1704-13. doi: 10.1016/j.ejca.2015.05.017. Epub 2015 Jun 3. PMID 26049686
- [Derived] Weeraratne D, Chen A, Pennucci JJ, Wu CY, Zhang K, Wright J, Perez-Ruixo JJ, Yang BB, Kaliyaperumal A, Gupta S, Swanson SJ, Chirmule N, Starcevic M. Immunogenicity of panitumumab in combination chemotherapy clinical trials. BMC Clin Pharmacol. 2011 Nov 9;11:17. doi: 10.1186/1472-6904-11-17. PMID 22070868
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 23 August 2006 and last patient enrolled 01 February 2008.
  Participant flow data are reported as of the data cut-off date of 28 August 2009.
Groups:
- FOLFOX + Panitumumab: Participants were randomized to panitumumab, 6 mg/kg on Day 1 and FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
- FOLFOX Alone: Participants were randomized to FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or until unacceptable toxicity.
Period: Overall Study
Arm/Group | FOLFOX + Panitumumab | FOLFOX Alone
Started | 593 | 590
Received Study Drug | 586 (One participant randomized to this group did not receive any panitumumab) | 583
Completed | 492 (Indicates participants who had completed the safety visit 30 days after last dose or had died) | 495 (Indicates participants who had completed the safety visit 30 days after last dose or had died)
Not Completed | 101 | 95
Not completed — Ineligibility determined | 4 | 2
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 13 | 18
Not completed — Physician Decision | 3 | 3
Not completed — Lost to Follow-up | 10 | 3
Not completed — Protocol-specified criteria | 6 | 6
Not completed — Other | 41 | 47
Not completed — Ongoing | 20 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFOX + Panitumumab | FOLFOX Alone | Total
Number analyzed (Participants) | 593 | 590 | 1183
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.1) | 60.3 (11.0) | 60.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 232 | 439
  Male | 386 | 358 | 744
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 530 | 540 | 1070
  Black or African American | 8 | 15 | 23
  Hispanic or Latino | 42 | 26 | 68
  Asian | 8 | 4 | 12
  Other | 5 | 5 | 10
Geographic Region [Number; unit: participants] — Stratification factor. Rest of world includes South America, eastern Europe, South Africa and Mexico
  participants
    Western Europe, Canada and Australia | 332 | 329 | 661
    Rest of world | 261 | 261 | 522
KRAS Status [Number; unit: participants] — KRAS, the human homolog of the Kirsten rat sarcoma-2 virus oncogene
  participants
    Wild-type KRAS | 325 | 331 | 656
    Mutant KRAS | 221 | 219 | 440
    Unevaluable KRAS | 47 | 40 | 87
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; Grade 3: Capable of only limited self care, confined to a bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; Grade 5: Dead
  participants
    Grade 0 | 332 | 320 | 652
    Grade 1 | 230 | 238 | 468
    Grade 2 | 31 | 29 | 60
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 1 | 1
    Mising/Unknown | 0 | 2 | 2
Primary tumor type [Number; unit: participants]
  Colon cancer | 394 | 398 | 792
  Rectal cancer | 199 | 192 | 391

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS), assessed by central radiological assessment, was defined as the time from randomization to disease progression per modified response evaluation criteria in solid tumors (RECIST) criteria or death. Participants who were alive but did not meet criteria for progression by the data cutoff date were censored at their last evaluable disease assessment date. Progressive disease is defined as a ≥ 20% increase in the size of target lesions or unequivocal progression of existing non-target lesions or any new lesions.
Time Frame: From randomization until the data cutoff date of 30 September 2008. Maximum follow-up time was 109 weeks.
Population: KRAS Efficacy Analysis Set (participants for whom KRAS status was assessed)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Wild-type KRAS - FOLFOX + Panitumumab: Participants with wild-type KRAS were randomized to panitumumab, 6 mg/kg on Day 1 and FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
- Wild-type KRAS - FOLFOX: Participants with wild-type KRAS were randomized to FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or until unacceptable toxicity.
- Mutant KRAS - FOLFOX + Panitumumab: Participants with mutant KRAS were randomized to panitumumab, 6 mg/kg on Day 1 and FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
- Mutant KRAS - FOLFOX: Participants with mutant KRAS were randomized to FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or until unacceptable toxicity.
Arm/Group | Wild-type KRAS - FOLFOX + Panitumumab | Wild-type KRAS - FOLFOX | Mutant KRAS - FOLFOX + Panitumumab | Mutant KRAS - FOLFOX
Number analyzed (Participants) | 325 | 331 | 221 | 219
months | 9.6 [9.2 to 11.1] | 8.0 [7.5 to 9.3] | 7.3 [6.3 to 8.0] | 8.8 [7.7 to 9.4]
Statistical Analysis 1: Comparison: Wild-type KRAS - FOLFOX + Panitumumab vs Wild-type KRAS - FOLFOX; PFS in the Wild-type KRAS Efficacy Analysis Set was compared at a significance level of 5%; Test type: Superiority or Other; p = 0.0234, Stratified log-rank test — P-value is based on a 2-sided log-rank test stratified by Region (Western Europe, Canada and Australia vs. Rest of World) and ECOG score (0 or 1 vs. 2); Normal score = -2.27 — A normal score <0 indicates fewer than expected events for the panitumumab plus FOLFOX arm and therefore a longer progression-free survival time
Statistical Analysis 2: Comparison: Mutant KRAS - FOLFOX + Panitumumab vs Mutant KRAS - FOLFOX; PFS in the Mutant KRAS Efficacy Analysis Set was compared at a significance level of 5% conditional on first demonstrating a significant treatment effect in PFS in the Wild-type KRAS Efficacy Analysis Set; Test type: Superiority or Other; p = 0.0227, Stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Normal score = 2.28 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Overall Survival
Description: The definition of overall survival is the time from randomization to death; participants who were alive at the analysis data cutoff were censored at their last contact date.
Time Frame: From randomization until the data cutoff date of 28 August 2009. Maximum time on follow-up was 153 weeks.
Population: KRAS Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - FOLFOX + Panitumumab | Wild-type KRAS - FOLFOX | Mutant KRAS - FOLFOX + Panitumumab | Mutant KRAS - FOLFOX
Number analyzed (Participants) | 325 | 331 | 221 | 219
months | 23.9 [20.3 to 28.3] | 19.7 [17.6 to 22.6] | 15.5 [13.1 to 17.6] | 19.3 [16.5 to 21.8]
Statistical Analysis 1: Comparison: Wild-type KRAS - FOLFOX + Panitumumab vs Wild-type KRAS - FOLFOX; Overall survival comparisons in the wild-type KRAS Efficacy Analysis Set was performed at a significance level of 4.99% conditional on a statistically significant difference for PFS in the Wild-type KRAS Efficacy Analysis Set; Test type: Superiority or Other; p = 0.0723, Stratified log-rank test — cP-value is based on a 2-sided log-rank test stratified by Region (Western Europe, Canada and Australia vs. Rest of World) and ECOG score (0 or 1 vs. 2); Normal score = -1.80 — A normal score <0 indicates fewer than expected events for the panitumumab plus FOLFOX arm and therefore a longer overall survival time
Statistical Analysis 2: Comparison: Mutant KRAS - FOLFOX + Panitumumab vs Mutant KRAS - FOLFOX; Overall survival comparisons in the mutant KRAS Efficacy Analysis Set was performed at an significance level of 4.99% conditional on a statistically significant difference for PFS in the Mutant KRAS Efficacy Analysis Set; Test type: Superiority or Other; p = 0.0678, Stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Normal score = 1.83 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Participants were evaluated for tumor response per the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria every 8 weeks until disease progression. Objective response by central radiological assessment was defined as the incidence of either a confirmed complete or partial response (CR or PR) while on the first-line treatment, as determined by blinded independent central review and confirmed no less than 4-weeks after the criteria for response are first met. CR: Disappearance of all target and non-target lesions and no new lesions. PR: At least a 30% decrease in the sum of the longest diameter of target lesions and no progression of non-target or no new lesions, or, disappearance of all target lesions and the persistence of ≥ 1 non-target lesion not qualifying for either CR or progressive disease. Participants without a post-baseline assessment were considered non-responders.
Time Frame: Every 8 weeks until disease progression up to the data cut-off date of 30 September 2008; Maximum follow-up time was 109 weeks.
Population: KRAS Evaluable Central Tumor Response Analysis Set (subset of participants with at least one uni-dimensionally measurable lesion per the modified RECIST criteria per blinded central radiology review).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS - FOLFOX + Panitumumab | Wild-type KRAS - FOLFOX | Mutant KRAS - FOLFOX + Panitumumab | Mutant KRAS - FOLFOX
Number analyzed (Participants) | 317 | 323 | 215 | 211
percentage of participants | 55.21 [49.55 to 60.77] | 47.68 [42.12 to 53.28] | 39.53 [32.95 to 46.41] | 40.28 [33.61 to 47.24]
Statistical Analysis 1: Comparison: Wild-type KRAS - FOLFOX + Panitumumab vs Wild-type KRAS - FOLFOX; Test type: Superiority or Other; p = 0.0684, Stratified exact test; Adjusted for geographic region and ECOG score; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.98 to 1.87] — The odds ratio is defined as the odds of having an objective response in the panitumumab plus arm relative to the odds on the FOLFOX alone arm
Statistical Analysis 2: Comparison: Mutant KRAS - FOLFOX + Panitumumab vs Mutant KRAS - FOLFOX; Test type: Superiority or Other; p = 0.9822, Stratified exact test; Adjusted for geographic region and ECOG score; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.65 to 1.47] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Time to Progression
Description: Time to progression was defined as time from randomization date to date of disease progression per the modified RECIST criteria.
Time Frame: From randomization until the data cut-off date of 30 September 2008; Maximum follow-up time was 109 weeks.
Population: KRAS Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - FOLFOX + Panitumumab | Wild-type KRAS - FOLFOX | Mutant KRAS - FOLFOX + Panitumumab | Mutant KRAS - FOLFOX
Number analyzed (Participants) | 325 | 331 | 221 | 219
months | 10.8 [9.4 to 12.4] | 9.2 [7.7 to 9.9] | 7.5 [7.2 to 8.9] | 9.0 [7.7 to 9.5]

5. Secondary Outcome: Duration of Response
Description: Duration of response was calculated only for those participants with a confirmed CR or PR, as the time from the first CR or PR (subsequently confirmed within no less than 4 weeks) to first observed disease progression per modified RECIST criteria, based on a blinded central review.
Time Frame: as for outcome 3
Population: KRAS Evaluable Central Tumor Response Analysis Set: Responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - FOLFOX + Panitumumab | Wild-type KRAS - FOLFOX | Mutant KRAS - FOLFOX + Panitumumab | Mutant KRAS - FOLFOX
Number analyzed (Participants) | 175 | 154 | 85 | 85
months | 11.1 [9.5 to 13.0] | 8.8 [7.8 to 9.7] | 7.4 [5.9 to 8.3] | 8.0 [6.5 to 9.5]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event (SAE) is defined as an AE that • is fatal • is life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • other significant medical hazard. The relationship of the adverse event to the study treatment was assessed by the Investigator by means of the question: "Is there a reasonable possibility that the event may have been caused by the study treatment?"
Time Frame: From randomization until the data cut-off date of 28 August 2009; Maximum time on follow-up was 153 weeks.
Population: Safety analysis set; One participant was randomized to 'Panitumumab Plus FOLFOX', but received 'FOLFOX Alone' so is counted in that group.
Measure: Number; unit: participants
Arm/Group | FOLFOX + Panitumumab | FOLFOX Alone
Number analyzed (Participants) | 585 | 584
participants
  Any adverse event | 583 | 579
  Serious adverse event | 262 | 198
  Leading to discontinuation of any study drug | 136 | 84
  Treatment-related adverse event (TRAE) | 581 | 565
  Serious treatment-related adverse event | 162 | 89
  TRAE leading to discontinuation of any study drug | 117 | 63

ADVERSE EVENTS:
Time Frame: The median treatment period was around 7.7 months in the Panitumumab arm, and around 6.7 months in the Chemo alone arm.
Description: One participant was randomized to 'Panitumumab Plus FOLFOX', but received 'FOLFOX Alone' so is counted in that group.
  The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency threshold in either treatment group.
Groups:
- Panitumumab Plus FOLFOX: Participants received panitumumab, 6 mg/kg on Day 1 and FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
- FOLFOX Alone: Participants received FOLFOX chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or until unacceptable toxicity.
Arm/Group | Panitumumab Plus FOLFOX | FOLFOX Alone
Serious Adverse Events (participants affected / at risk) | 262/585 | 198/584
Other Adverse Events (participants affected / at risk) | 577/585 | 571/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFOX (N=585) | FOLFOX Alone (N=584)
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 14
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 10
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 10
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Anal erosion (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 58 | 17
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faecalith (Gastrointestinal disorders) | 1 | 0
Gastric dilatation (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 6 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 18 | 12
Intestinal perforation (Gastrointestinal disorders) | 3 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 3
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Retroperitoneal oedema (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 0
Subileus (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 18 | 12
Asthenia (General disorders) | 6 | 2
Catheter related complication (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter thrombosis (General disorders) | 0 | 3
Chest pain (General disorders) | 4 | 0
Chills (General disorders) | 0 | 3
Fatigue (General disorders) | 5 | 1
General physical health deterioration (General disorders) | 7 | 2
Hyperpyrexia (General disorders) | 1 | 0
Inflammation of wound (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 6 | 2
Multi-organ failure (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pelvic mass (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 2
Pyrexia (General disorders) | 16 | 15
Sudden death (General disorders) | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 2 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 4 | 4
Abdominal abscess (Infections and infestations) | 2 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Acne pustular (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 2
Biliary abscess (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 6 | 4
Catheter sepsis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 0
Central line infection (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Groin abscess (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 8
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 12 | 7
Septic shock (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 5
Urinary tract infection viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 2
Anal injury (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 3
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood culture positive (Investigations) | 1 | 0
Cardiac enzymes increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 20 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour local invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 2
Dysarthria (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 1
Personality disorder (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 8 | 6
Renal failure acute (Renal and urinary disorders) | 3 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 10 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter placement (Surgical and medical procedures) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 9 | 5
Embolism (Vascular disorders) | 1 | 1
Embolism venous (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 2
Iliac artery embolism (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 2 | 0
Venous thrombosis limb (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFOX (N=585) | FOLFOX Alone (N=584)
Anaemia (Blood and lymphatic system disorders) | 84 | 81
Leukopenia (Blood and lymphatic system disorders) | 48 | 50
Neutropenia (Blood and lymphatic system disorders) | 315 | 353
Thrombocytopenia (Blood and lymphatic system disorders) | 115 | 157
Conjunctivitis (Eye disorders) | 103 | 20
Lacrimation increased (Eye disorders) | 26 | 40
Abdominal pain (Gastrointestinal disorders) | 156 | 133
Abdominal pain upper (Gastrointestinal disorders) | 49 | 55
Constipation (Gastrointestinal disorders) | 154 | 155
Diarrhoea (Gastrointestinal disorders) | 349 | 282
Dry mouth (Gastrointestinal disorders) | 31 | 17
Dyspepsia (Gastrointestinal disorders) | 64 | 63
Nausea (Gastrointestinal disorders) | 261 | 287
Stomatitis (Gastrointestinal disorders) | 138 | 77
Vomiting (Gastrointestinal disorders) | 175 | 182
Asthenia (General disorders) | 132 | 117
Fatigue (General disorders) | 199 | 197
Mucosal inflammation (General disorders) | 143 | 87
Oedema peripheral (General disorders) | 61 | 47
Pyrexia (General disorders) | 170 | 149
Nasopharyngitis (Infections and infestations) | 31 | 25
Paronychia (Infections and infestations) | 120 | 0
Urinary tract infection (Infections and infestations) | 35 | 31
Weight decreased (Investigations) | 97 | 39
Anorexia (Metabolism and nutrition disorders) | 199 | 133
Dehydration (Metabolism and nutrition disorders) | 32 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 30 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 116 | 73
Hypomagnesaemia (Metabolism and nutrition disorders) | 175 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 67 | 68
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 39
Dizziness (Nervous system disorders) | 38 | 39
Dysaesthesia (Nervous system disorders) | 33 | 50
Dysgeusia (Nervous system disorders) | 77 | 79
Headache (Nervous system disorders) | 37 | 72
Lethargy (Nervous system disorders) | 24 | 30
Neuropathy peripheral (Nervous system disorders) | 110 | 138
Paraesthesia (Nervous system disorders) | 180 | 204
Peripheral sensory neuropathy (Nervous system disorders) | 77 | 89
Anxiety (Psychiatric disorders) | 44 | 31
Depression (Psychiatric disorders) | 34 | 25
Insomnia (Psychiatric disorders) | 80 | 82
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 84
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 79 | 53
Acne (Skin and subcutaneous tissue disorders) | 74 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 80 | 56
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 188 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 120 | 20
Erythema (Skin and subcutaneous tissue disorders) | 94 | 22
Nail disorder (Skin and subcutaneous tissue disorders) | 49 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 55 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 128 | 26
Rash (Skin and subcutaneous tissue disorders) | 305 | 39
Skin fissures (Skin and subcutaneous tissue disorders) | 89 | 2
Hypertension (Vascular disorders) | 26 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.